CLINICAL TRIAL: NCT00448994
Title: Serial Monitoring of Adenovirus and Fungal Load by Real-Time, Quantitative Polymerase Chain Reaction (PCR) Assay and Correlation With Outcomes in Pediatric Hematopoietic Stem Cell Transplant Patients
Brief Title: Adenovirus and Fungal Load in Pediatric Stem Cell Transplant Patients
Status: Withdrawn | Type: Observational
Why Stopped: Method development/validation
Sponsor: Steven B. Kleiboeker (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Steven B. Kleiboeker, VP, Scientific Affairs, ViraCor Laboratories
Organization: ViraCor Laboratories (Industry)
Other Study IDs: 05-0101
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Adenovirus; Other Mycoses
Keywords: adenovirus, fungal, diagnostics, children
MeSH Terms: conditions — Adenoviridae Infections

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is designed to determine the rate at which stem cell transplant patients can develop infection caused by a group of viruses, known as adenovirus, and common fungi. Stem cells are unspecialized cells, capable of producing more stem cells or other specialized cells, and are used to replace damaged or diseased cells. The study will be conducted in children (2-17years old) being transplanted with stem cells from a donor. Patients undergoing stem cell transplantation are more likely to develop infections as their immune systems are weakened. Blood, stool, urine and throat swab samples will be collected (for at least 100 days on a weekly basis) to detect infection(s) caused by adenovirus or fungus. Subjects will participate for up to 1 year following the transplant procedure.

DETAILED DESCRIPTION:
This study is a multi-center observational study to determine the usefulness of real time PCR in the detection of adenovirus and fungal infections in patients following HSCT. Quantitative viral load monitoring will be evaluated to establish correlation with clinical symptoms and to measure the effectiveness of the therapeutic interventions. Samples will be collected prior to HSCT and on a scheduled weekly basis for 100 days post-HSCT and after that when patients show signs of infection. Patients' signs and symptoms and outcomes will be recorded for correlation with viral load. In addition, viral cultures will be performed on the same schedule as PCR assay using 3 samples (throat swab, stool, and urine). The study will be conducted at approximately 6 centers in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients greater than or equal to 2 years of age.
2. Allogeneic HSCT.
3. Willing and able to give signed informed consent, or have a legally authorized representative who is willing to give consent. Informed assent will be required for children <18 years of age.
4. Reliable and willing to make themselves available for the duration of the study.

Exclusion Criteria:

1. Autologous transplant patients are not eligible for the study.
2. Patients previously enrolled in the study may not reenroll in the event of a subsequent HSCT.
3. Pediatric patients less than 2 years of age are not eligible for the study.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Method development | 3 years

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Mercy Hospital, Kansas City, Missouri
  - Texas Transplant Institute, San Antonio, Texas